CLINICAL TRIAL: NCT01437319
Title: Mucin Balls and Corneal Inflammation Events
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CR-005016
Record Dates: First submitted 2011-09-16; First posted 2011-09-20 (Estimated); Results first posted 2016-02-25 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2016-01

CONDITIONS: Corneal Inflammation; Corneal Infiltrative Events
MeSH Terms: conditions — Keratitis

ARMS (2):
- lotrafilcon A, comfilcon A (Active Comparator): All subjects are assigned to lotrafilcon A during a run-in (Phase 1) and then randomized to one of two lenses. This arm is assigned to comfilcon A at phase 2. Subjects classified as a Neophyte wore etafilcon A for 2-weeks before entering the run-in period in Phase I.
  Interventions: Device: lotrafilcon A; Device: comfilcon A; Other: etafilcon A
- lotrafilcon A, balafilcon A (Active Comparator): All subjects are assigned to lotrafilcon A during a run-in (Phase 1) and then randomized to one of two lenses. This arm is assigned to balafilcon A at phase 2. Subjects classified as a Neophyte wore etafilcon A for 2-weeks before entering the run-in period in Phase I.
  Interventions: Device: lotrafilcon A; Device: balafilcon A; Other: etafilcon A

INTERVENTIONS:
Device: lotrafilcon A — To be used during run-in phase only.
Device: comfilcon A — To be assigned at randomization at phase 2 only.
  Arms: lotrafilcon A, comfilcon A
Device: balafilcon A — To be assigned at randomization during phase 2 only.
  Arms: lotrafilcon A, balafilcon A
Other: etafilcon A — Assigned to Neophytes during Phase I for a 2-week period

SUMMARY:
The purpose of this study is to determine if the formation of mucin balls is a marker for protection from inflammatory events to the cornea and if mucin balls play a role in protection during extended contact lens wear.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years
* Free of any active anterior segment disorders that would preclude safe contact lens wear. Active anterior segment disorders and evidence of central microbial keratitis (via a large, >1mm central deep stromal scar) are not allowed. However, evidence of past Contact Lens-Induces Peripheral Ulcer (CLPU) will be allowed so long as no more then three such scars are detected bilaterally. Evidence of more than 3 CLPU-like scars places excessive risk on the subject for a subsequent Corneal Infiltrate Event (CIE).
* Correctable vision to 20/25 or better in each eye with spectacles. Amblyopia will be excluded.
* Flat and steep corneal curvatures from keratometry readings must be between 39.00 and 48.50 D, respectively.
* Own or agree to purchase a pair of spectacles that can be worn when lenses are removed or in cases of ocular discomfort or emergency.
* Correctable vision to 20/30 or better at distance with dispensed contact lenses.

Exclusion Criteria:

* Use/wear of rigid gas permeable lenses within the last 30 days or Poly (methyl methacrylate) (PMMA) lenses within the last 3 months.
* Immunocompromising disease or insulin dependent diabetes or any other systemic disease that in the investigator's opinion will affect ocular health or increase risk during extended wear.
* Chronic use of systemic corticosteroids (with the exception of corticosteroid inhalers) or any other medication that in the investigator's opinion will affect ocular physiology or study participation.
* Ocular disease or condition such as aphakia, corneal dystrophies, corneal edema, external ocular infection, iritis, or had any anterior segment surgery.
* Use of any ocular medications in the last 2 weeks.
* Less than or equal to grade 2 on any of the slit lamp observations of: upper tarsal papilla, corneal staining, corneal neovascularization, conjunctival injection, and lid erythema or scales.
* Currently pregnant or lactating.
* Smoker
* Swimming routine of more than twice per month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 289 (Actual)
Dates: Start 2011-09; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Beachwood, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio

REFERENCES:
- [Derived] Szczotka-Flynn LB, Jiang Y, Stiegemeier MJ, Mutti DO, Walline J, Wilson T, Debanne S; Mucin Ball Study Group. Mucin Balls Influence Corneal Infiltrative Events. Optom Vis Sci. 2017 Apr;94(4):448-457. doi: 10.1097/OPX.0000000000001045. PMID 28195933

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 289 Subjects were enrolled in the study. 7 subjects did not meet the eligibility criteria. 282 subjects entered Phase I. During Phase I, 55 subjects were either lost to follow-up or discontinued. The remaining 227 subjects were randomized to either comfilcon A or balafilcon A and entered Phase II. 146 subjects completed Phase II
Pre-assignment Details: During Phase I, subjects are classified as either repeated Mucin Ball former or Non-Repeat Mucin Ball former. The 227 subjects that entered Phase II kept there Mucin ball classification, but were still randomized to either comfilcon A or balafilcon A. All comparisons are made between Mucin Ball classification
Groups:
- Lotrafilcon A: All subjects received lotrafilcon A in Phase I.
- Comfilcon A: Subjects that received comfilcon A lens in Phase II.
- Balfilcon A: Subjects that received balafilcon A lens in Phase II.
Period: Phase I
Arm/Group | Lotrafilcon A | Comfilcon A | Balfilcon A
Started | 282 | 0 | 0
Completed | 227 | 0 | 0
Not Completed | 55 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Study related symptoms/complaints | 27 | 0 | 0
Not completed — Withdrawal by Subject | 25 | 0 | 0
Period: Phase II
Arm/Group | Lotrafilcon A | Comfilcon A | Balfilcon A
Started | 0 | 115 | 112
Completed | 0 | 71 | 75
Not Completed | 0 | 44 | 37
Not completed — Withdrawal by Subject | 0 | 8 | 16
Not completed — Lost to Follow-up | 0 | 7 | 2
Not completed — Study related symptoms/complaints | 0 | 28 | 19
Not completed — Protocol Violation | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The analysis population consists of all subjects that entered Phase 1.
Groups:
- Overall: The analysis population consists of all subjects that were enrolled into the study.
Arm/Group | Overall
Number analyzed (Participants) | 282
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.8 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 182
  Male | 100
Region of Enrollment [Number; unit: participants]
  United States | 282

OUTCOME MEASURES:

1. Primary Outcome: Corneal Infiltrate Events - Phase I
Description: The percentage of Subjects that experienced Corneal Inflammatory Events within their Mucin Ball classification.
Time Frame: 1-Month Follow-up
Population: The analysis population consists of subjects that completed all study visits in Phase I without a major protocol deviation and were correctly classified as either repeat Mucin Ball former or Non-repeat Mucin Ball former. Five subjects had incorrect Mucin Ball classification and 8 subjects met study objective.
Measure: Number; unit: percentage of subjects
Groups:
- Repeat Mucin Ball Former: Subjects that were classified as being repeat Mucin Ball former.
- Non-repeat Mucin Ball Former: Subjects that were classified as Non-repeat Mucin Ball Former.
Arm/Group | Repeat Mucin Ball Former | Non-repeat Mucin Ball Former
Number analyzed (Participants) | 161 | 53
percentage of subjects | 18.6 | 5.7

2. Primary Outcome: Corneal Infiltrate Event- Phase II
Description: The percentage of Subjects that experienced Corneal Inflammatory Events within their Mucin Ball classification.
Time Frame: 12-Month Follow-up
Population: The analysis population consists of subjects that were enrolled into Phase II and were correctly classified as either repeat Mucin Ball former or Non-repeat Mucin Ball former. Twenty- three subjects had incorrect Mucin ball classification.
Measure: Number; unit: percentage of subjects
Arm/Group | Repeat Mucin Ball Former | Non-repeat Mucin Ball Former
Number analyzed (Participants) | 153 | 43
percentage of subjects
  balafilcon A, N=66, N=28 | 4.5 | 3.6
  comfilcon A, N=87, N=15 | 14.9 | 33.3

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Comfilcon A: Subjects who received comfilcon A in Phase II of the study.
- Balafilcon A: Subjects who received balafilcon A in Phase II of the study
- Lotrafilcon A: All Subjects received lotrafilcon A in Phase I of the study.
Arm/Group | Comfilcon A | Balafilcon A | Lotrafilcon A
Serious Adverse Events (participants affected / at risk) | 0/115 | 0/112 | 0/282
Other Adverse Events (participants affected / at risk) | 30/115 | 24/112 | 23/282
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Comfilcon A (N=115) | Balafilcon A (N=112) | Lotrafilcon A (N=282)
Asymptomatic corneal scar (Eye disorders) | 6/114 (6) | 3 (3) | 3 (3)
Cornea Lens Peripheral Ulcer (CLPU) (Eye disorders) | 12 (13) | 3 (3) | 10 (10)
Conjunctivitis (Eye disorders) | 12 (25) | 12 (21) | 8 (12) — Includes Contact lens papillary, viral, bacterial, and allergic
SEALs (Eye disorders) | 0 (0) | 6 (6) | 2 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days